CLINICAL TRIAL: NCT01134965
Title: An Open Two-way Cross-over Study to Evaluate the Effect of Multiple Doses of Flibanserin 100 mg Film-coated Tablets Given Once Daily on the Single Dose Pharmacokinetics of Digoxin 0.5 mg in Healthy Male and Female Volunteers
Brief Title: to Evaluate Effect of Multi Doses Flibans 100 mg Film-c Tablets on Single Dose PK of Digoxin 0.5 mg, Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 511.158; 2010-018950-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
MeSH Terms: interventions — flibanserin; Digoxin

ARMS (2):
- Digoxin plus Flibanserin (Experimental): Flibanserin 100 mg tablets once daily for 7 days plus Digoxin 0.5 mg (2 tables of 0.25 mg) as single dose
  Interventions: Drug: Flibanserin plus Digoxin
- Digoxin (Experimental): Digoxin 0.5 mg as single dose
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Flibanserin plus Digoxin — Flibanserin 100 mg once daily for 7 days plus Digoxin 0.5 mg as single dose
  Arms: Digoxin plus Flibanserin
Drug: Digoxin — Digoxin 0.5 mg as single dose
  Arms: Digoxin

SUMMARY:
The aim of this trial is to investigate the effect of multiple doses of flibanserin on the single dose pharmacokinetics of digoxin in healthy female and male volunteers. Digoxin is a narrow therapeutic index drug for which a large number of relevant drug-drug interactions are known. Flibanserin is now under evaluation in postmenopausal women which increases the likelihood that flibanserin and digoxin will be administered together in the clinical setting.

ELIGIBILITY:
Inclusion criteria:

healthy male and female subjects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of digoxin in plasma after single dose (Cmax) | 72 hours
Area under the concentration-time curve of digoxin in plasma over the time interval 0 to infinity (AUC0-inf) | 72 hours

SECONDARY OUTCOMES:
Renal clearance of digoxin from time 0 to 24 hours after drug administration (CLR,0-24) | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 511.158.1 Boehringer Ingelheim Investigational Site, Biberach, Germany